CLINICAL TRIAL: NCT04985032
Title: Accelerated Partial Breast Irradiation (APBI) Using Stereotactic Body Radiation Therapy (SBRT): a Multicenter, Observational Clinical Trial
Brief Title: Accelerated Partial Breast Irradiation (APBI) Using Stereotactic Body Radiation Therapy (SBRT)
Status: Recruiting | Type: Observational
Sponsor: RPCR, Inc. (Other)
Collaborators: CyberKnife Coalition (Unknown)
Responsible Party: Sponsor
Other Study IDs: RPCR-breast 01
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Ductal Carcinoma in Situ; Invasive Ductal Carcinoma of Female Breast
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Treatment technique used to deliver a highly focused and accurate radiation dose to a defined target volume outside the brain; the entire course of therapy delivered in five fractions or less

SUMMARY:
This is a multi-institutional, prospective, observational registry investigating the safety and efficacy of Accelerated Partial Breast Irradiation (APBI) using a Stereotactic Body Radiation Therapy (SBRT) delivery technique that incorporates real-time image guidance, noncoplanar fields, and respiratory tracking. The study will accrue 200 patients who will be treated to a dose of 30 Gy over the course of 5 fractions. These subjects will then have a follow up time of 5 years

DETAILED DESCRIPTION:
RADIATION TREATMENT GUIDELINES and DOSIMETRY Fiducial Placement Prior to enrollment, patients will undergo breast conservation surgery preferably with fiducial markers implanted at the time of surgery or under ultrasonic guidance25

Patients treated with gantry-based SBRT preferably will have fiducials placed at the time of surgery.

For patients being treated with CyberKnife SBRT, four gold markers will be placed intraoperatively or ultrasonically to define the superior, inferior, medial, and lateral boundaries of the lumpectomy cavity in accordance with the manufacturer's (Accuray) documentation. At least three fiducials will be required for target tracking purposes to allow for rotational changes.

Simulation Linear Accelerator SBRT For treatments on a gantry-based linear accelerator, patients will be positioned supine with the arms elevated. CT scans will be obtained with 1.25 mm thickness and will be acquired with free breathing as well as additional scans as needed for motion control or gating. 4DCT, MRI and PET imaging may be used to assist in determining motion estimation.

CyberKnife SBRT For treatment on a robotic system, a contrast enhanced CT simulation is to be performed with 1 mm slices with the patient's arms at her sides in the supine position. The scan is to be performed with end-inspiratory breath hold from the thyroid to below the lungs. Breast immobilization devices including a vacuum mattress and a bra system will be allowed however bolus should not be used. Fiducial tracking (Synchrony) is to be used for motion tracking.

DOSIMETRY Target and Organs at Risk (OAR) contours

The following structures are to be contoured in all patients:

Tumor cavity (GTV) as defined on CT including all fiducials implanted on CT images Clinical Target Volume (CTV) defined as the tumor cavity expanded by a uniform 15 mm margin. The CTV will not extend beyond the skin, breast or chestwall Planning Tumor Volume (PTV) for SBRT will be defined as the CTV plus 3 - 5 mm as needed at the treating physician's discretion. PTV will be limited to GTV plus 20 mm margin Skin is defined as <5 mm inside the external contour Chest wall includes the ribs and intercoastal musculature but does not include the pectoralis Heart contour begins below the level of where the pulmonary trunk branches into the left and right pulmonary arteries Lungs are to be contoured separately Spinal canal Breasts are to be contoured separately Dose Prescription The total prescribed dose to the PTV is 30 Gy delivered in 5 equal fractions of 6 Gy per day delivered on alternating days over 5 -10 total days. The prescribed dose must cover at least 95% of the PTV.

ELIGIBILITY:
Inclusion Criteria:

1. Women 50 years or older
2. Low to intermediate grade DCIS or invasive ductal carcinoma
3. Tumor size < 2 cm invasive ductal carcinoma and < 2.5 cm DCIS
4. Well defined lumpectomy cavity on CT
5. Clear surgical ink margins > 2mm for invasive cancer and > 3 mm for DCIS
6. Node negative
7. Unifocal lesion
8. ER and/or PR positive
9. HER-2 negative
10. BRCA negative
11. Lumpectomy cavity must be < 30% of whole breast volume

Exclusion Criteria:

1. Lobular histology
2. Angiolymphatic invasion
3. Multiple foci of disease
4. Lymphovascular invasion
5. Active lupus or sarcoid
6. Distant metastases
7. Non-epithelial malignancies
8. Synchronous contralateral breast cancer
9. Grade 2 or higher oncoplastic surgery
10. Ipsilateral pacemaker
11. Ipsilateral breast implant
12. Neoadjuvant chemotherapy
13. Prior ipsilateral breast cancer or thoracic radiation
14. Poor breast integrity
15. Paget's Disease of the nipple
16. Pregnant patients
17. Severe cardiac, pulmonary, or liver diseases

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SBRT for treatment of the surgical cavity following partial mastectomy for women with early-stage breast cancer will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Breast Cosmesis as measured by NRG-Radiation Therapy Oncology Group (RTOG) global cosmetic score (GCS) and the Harvard Cosmesis Scale (HCS) | 2-3 years
  physician and patient assessment of breast cosmetic result following SBRT
Acute breast toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 1-6 weeks
  assessment of skin and breast tissue changes during and immediately following SBRT
Other late toxicities as measured by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 3-60 months
  assessment of pulmonary, cardiac and chest wall changes following SBRT

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CyberKnife Center of South Florida in Stuart, Stuart, Florida
  - CyberKnife Centers of Tampa Bay, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Comprehensive Cancer Network. Invasive Breast Cancer (Version 1.2021) https://www.nccn.org/professionals/physician_gls/pdf/breast.pdf
- [Background] 2Bonfantini F, De Martin E, Giandini T, Fumagalli ML, Cavallo A, Pinzi V, et al. A Dosimetric Comparison between Three Different External Photon Beam Techniques for Accelerated Partial Breast Irradiation. Clin Oncol. 2018; 3:1501.
- [Background] Hepel JT, Tokita M, MacAusland SG, Evans SB, Hiatt JR, Price LL, DiPetrillo T, Wazer DE. Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1290-6. doi: 10.1016/j.ijrobp.2009.01.009. Epub 2009 Apr 22. PMID 19395195
- [Background] Wolmark N, Curran WJ, Vicini F, White J, Costantino JP, Arthur D, Kuske R, Rabinovitch R, Julian TB, Parda DS. Response to "Unacceptable cosmesis in a protocol investigating intensity-modulated radiotherapy with active breathing control for accelerated partial-breast irradiation" (Int J Radiat Oncol Biol Phys 2010;76:71-78) and "Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation" Int J Radiat Oncol Biol Phys 2009;75:1290-1296). Int J Radiat Oncol Biol Phys. 2010 May 1;77(1):317; author reply 318. doi: 10.1016/j.ijrobp.2009.12.033. No abstract available. PMID 20394863
- [Background] Whelan TJ, Julian JA, Berrang TS, Kim DH, Germain I, Nichol AM, Akra M, Lavertu S, Germain F, Fyles A, Trotter T, Perera FE, Balkwill S, Chafe S, McGowan T, Muanza T, Beckham WA, Chua BH, Gu CS, Levine MN, Olivotto IA; RAPID Trial Investigators. External beam accelerated partial breast irradiation versus whole breast irradiation after breast conserving surgery in women with ductal carcinoma in situ and node-negative breast cancer (RAPID): a randomised controlled trial. Lancet. 2019 Dec 14;394(10215):2165-2172. doi: 10.1016/S0140-6736(19)32515-2. Epub 2019 Dec 5. PMID 31813635
- [Background] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636
- [Background] 7White J. Cosmetic Outcomes from Post Lumpectomy Whole Breast Irradiation (WBI) Versus Partial Breast Irradiation (PBI) on the NRG Oncology/NSABP B39-RTOG 0413 Phase III Clinical Trial. ASTRO Annual Meeting. November 10, 2019.
- [Background] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Background] Meattini I, Marrazzo L, Saieva C, Desideri I, Scotti V, Simontacchi G, Bonomo P, Greto D, Mangoni M, Scoccianti S, Lucidi S, Paoletti L, Fambrini M, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Pallotta S, Livi L. Accelerated Partial-Breast Irradiation Compared With Whole-Breast Irradiation for Early Breast Cancer: Long-Term Results of the Randomized Phase III APBI-IMRT-Florence Trial. J Clin Oncol. 2020 Dec 10;38(35):4175-4183. doi: 10.1200/JCO.20.00650. Epub 2020 Aug 24. PMID 32840419
- [Background] Hoekstra N, Habraken S, Swaak-Kragten A, Breedveld S, Pignol JP, Hoogeman M. Reducing the Risk of Secondary Lung Cancer in Treatment Planning of Accelerated Partial Breast Irradiation. Front Oncol. 2020 Aug 18;10:1445. doi: 10.3389/fonc.2020.01445. eCollection 2020. PMID 33014782
- [Background] Rahimi A, Thomas K, Spangler A, Rao R, Leitch M, Wooldridge R, Rivers A, Seiler S, Albuquerque K, Stevenson S, Goudreau S, Garwood D, Haley B, Euhus D, Heinzerling J, Ding C, Gao A, Ahn C, Timmerman R. Preliminary Results of a Phase 1 Dose-Escalation Trial for Early-Stage Breast Cancer Using 5-Fraction Stereotactic Body Radiation Therapy for Partial-Breast Irradiation. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):196-205.e2. doi: 10.1016/j.ijrobp.2017.01.020. Epub 2017 Jan 12. PMID 28586960
- [Background] Rahimi A, Morgan HE, Kim DW, Zhang Y, Leitch M, Wooldridge R, Goudreau S, Haley B, Rao R, Rivers A, Spangler AE, Jones RT, Stevenson S, Staley J, Albuquerque K, Ahn C, Neufeld S, Alluri PG, Ding C, Garwood D, Seiler S, Zhao B, Gu X, Timmerman R. Cosmetic Outcomes of a Phase 1 Dose Escalation Study of 5-Fraction Stereotactic Partial Breast Irradiation for Early Stage Breast Cancer. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):772-782. doi: 10.1016/j.ijrobp.2021.01.015. Epub 2021 Jan 18. PMID 33476737